CLINICAL TRIAL: NCT04103060
Title: A Phase 2a, Randomized, Double-Blind, Vehicle-Controlled Study to Assess the Safety, Tolerability, and Systemic Exposure of Cerdulatinib Gel, 0.37% in Adults With Vitiligo
Brief Title: Safety and Tolerability Study of Cerdulatinib Gel, 0.37% in Adults With Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermavant Sciences GmbH (Industry)
Responsible Party: Sponsor
Organization: Dermavant Sciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMVT-502-2101
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — 4-(cyclopropylamino)-2-((4-(4-(ethylsulfonyl)piperazin-1-yl)phenyl)amino)pyrimidine-5-carboxamide; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cerdulatinib 0.37% gel (Experimental): Cerdulatinib 0.37% gel applied topically twice daily
  Interventions: Drug: Cerdulatinib 0.37% gel
- Vehicle gel (Placebo Comparator): Vehicle gel applied topically twice daily
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: Cerdulatinib 0.37% gel — Cerdulatinib 0.37% gel applied topically twice daily for 6 weeks
  Other Names: DMVT-502
  Arms: Cerdulatinib 0.37% gel
Drug: Vehicle gel — Vehicle gel applied topically twice daily for 6 weeks
  Arms: Vehicle gel

SUMMARY:
This is a phase 2a, randomized, double-blind, vehicle-controlled study to assess the safety, tolerability, and systemic exposure of cerdulatinib gel, 0.37% in adults with vitiligo

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 18 and older with a confirmed clinical diagnosis of vitiligo for at least 3 months, including ≥0.5% to ≤30% BSA involvement.
* Females of child bearing potential and male subjects who are engaging in sexual activity that could lead to pregnancy agree to follow the specified contraceptive guidance throughout the study
* Capable of giving informed consent

Exclusion Criteria:

* Diagnosis of segmental vitiligo
* Subjects with concurrent conditions or history of other diseases (e.g., current or chronic history of liver disease) that could affect the safety of the subject or the implementation of this study
* Use of any prohibited medication within the indicated period before the first dose of study drug
* Pregnant or lactating females
* Ultraviolet (UV) light therapy or prolonged exposure to natural or artificial sources of UV radiation within 8 weeks prior to the Baseline visit and/or plans to have such exposures during the study which could potentially impact the subject's vitiligo
* The subject has received an investigational product within the following time period prior to the first dosing day: 4 weeks or 5 half-lives (whichever is longer).
* Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular (CV) system abnormalities or laboratory test value abnormality that will affect the health of the subject or interfere with interpretation of the results
* History of sensitivity to the study drug, or components thereof or a history of drug or other allergy that contraindicates the subject's participation in the study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Vital signs | Baseline through Week 7
  Body temperature, blood pressure, pulse (heart rate), and breathing rate (respiratory rate)
Laboratory Values | Baseline through Week 7
  Clinically significant abnormal lab values
Adverse Events | Baseline through Week 7
  Frequency, severity, and duration of adverse events
Local Tolerability Scale Score | Baseline, Week 2, Week 4, Week 6, and Week 7
  Assessment of local site investigational product administration

SECONDARY OUTCOMES:
Concentration of cerdulatinib | Days 1, 15, 29 and 43
  Plasma concentration
Blister fluid biomarker concentration | Baseline and Week 6
  From active treated lesions and untreated nonlesional skin

CONTACTS AND LOCATIONS:
Overall Officials: Michael McLaughlin, Study Director — Dermavant Sciences GmbH
Locations (2):
- United States (2):
  - Dermavant Investigational Site, Irvine, California
  - Dermavant Investigational Site, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No